CLINICAL TRIAL: NCT02887859
Title: A Phase 2 Study for the Evaluation of Safety and Efficacy of Humacyte's Human Acellular Vessel for Use as a Vascular Prosthesis for Femoro-Popliteal Bypass in Patients With Peripheral Arterial Disease
Brief Title: Humacyte's HAV for Femoro-Popliteal Bypass in Patients With PAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Humacyte, Inc. (Industry)
Collaborators: Atlantic Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-PRO-V004
Record Dates: First submitted 2016-08-25; First posted 2016-09-02 (Estimated); Results first posted 2023-12-19 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HAV Treatment (Experimental): Human Acellular Vessel (HAV)
  Interventions: Biological: Human Acellular Vessel (HAV)

INTERVENTIONS:
Biological: Human Acellular Vessel (HAV) — Patients will be implanted with a Human Acellular Vessel (HAV) as a femoro-popliteal bypass conduit using standard vascular surgical techniques

SUMMARY:
This study will evaluate how well Humacyte's Human Acellular Vessel (HAV) works when surgically implanted into a leg to improve blood flow in patients with peripheral arterial disease (PAD). This study will also evaluate how safe it is to use the HAV in this manner.

DETAILED DESCRIPTION:
This is a prospective, open label, single treatment arm, multicenter phase 2 study to evaluate the safety and efficacy of the HAV in patients with PAD undergoing femoro-popliteal bypass surgery. The primary objective of this study is to evaluate the safety and tolerability of the HAV in these patients and to determine the patency of the Humacyte HAV at 12 months post-implantation. The secondary objectives of this study are to further assess safety in terms of PRA response, and to determine the rates of HAV interventions required to keep the HAV patent. There is no formal hypothesis testing planned; the study involves only a single, open-label treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with disabling symptomatic peripheral arterial disease

   1. Rutherford stage 4 or 5 who require femoro-popliteal bypass surgery or
   2. Rutherford stage 3 with severe claudication (less than 50 yards AND causing severe impairment of ability to work or undertake social activities)
2. Ankle - brachial index ≤ 0.6 in the study leg
3. Patient has failed adequate medical therapy which included

   1. Exercise program
   2. Smoking cessation therapy
   3. Control of diabetes, hypertension and dyslipidemias
   4. Antiplatelet therapy
4. Preoperative angiography or CT angiography shows superficial femoral artery occlusion AND required Humacyte Human Acellular Vessel (HAV) length of ≤ 38cm. This imaging may have been conducted up to 6 months prior to study entry provided that the patient's symptoms have remained stable since that time
5. Preoperative imaging shows at least one below knee vessel patent to the ankle with good runoff
6. Proximal HAV anastomosis is expected to be to the common femoral artery below the inguinal ligament or to the superficial femoral artery
7. Distal anastomosis is expected to be to the popliteal artery above the knee
8. Femoral artery occlusion is not considered suitable for endovascular treatment; e.g. long segment chronic total occlusion, previous failed stent or stent graft in the superficial femoral artery, previous failed endovascular treatment where the lesion could not be crossed
9. Autologous vein graft is not feasible in the judgment of the treating surgeon; e.g. because all suitable veins have been used previously for coronary or peripheral bypass, or pre-operative vein mapping shows inadequate length or quality of vein to complete the planned bypass
10. Aged 18 to 85 years old, inclusive
11. Hemoglobin ≥ 10g/dL and platelet count ≥ 100,000/mm3 at screening
12. Other hematological and biochemical parameters within a range considered acceptable for the administration of general anesthesia at screening
13. Adequate liver function, defined as serum bilirubin ≤ 1.5 mg/dL; and INR ≤ 1.5 at screening
14. Able to communicate meaningfully with investigative staff, competent to give written informed consent, and able to comply with entire study procedures
15. Life expectancy of at least 1 year

Exclusion Criteria:

1. Leg at high risk of amputation (SVS WIfI stage 4)
2. Recent clinically significant trauma to the leg receiving the HAV
3. Severe active infection (SVS foot infection grade 3) in the leg receiving the HAV
4. Distal anastomosis planned to a below knee artery
5. History or evidence of severe cardiac disease (NYHA Functional Class III or IV), myocardial infarction within six months prior to study entry (Day 1), ventricular tachyarrhythmias requiring continuing treatment, or unstable angina
6. Stroke within six (6) months prior to study entry (Day 1)
7. Chronic renal disease such that multiple administrations of contrast agents may pose an increased risk of nephrotoxicity (eGFR<45mL/min)
8. Uncontrolled diabetes (HbA1c >10% at screening)
9. Treatment with any investigational drug or device within 60 days prior to study entry (Day 1)
10. Cancer that is being actively treated with a cytotoxic agent
11. AIDS / HIV infection
12. Documented hypercoagulable state or history as defined as either:

    1. a biochemical diagnosis (e.g. Factor V Leiden, Protein C deficiency, etc.) - OR -
    2. a clinical history of thrombophilia as diagnosed by 2 or more spontaneous intravascular thrombotic events (e.g. DVT, PE, etc.) within the previous 5 years
13. Spontaneous or unexplained bleeding diathesis clinically documented within the last 5 years or a biochemical diagnosis (e.g. von Willebrand disease, etc.).
14. Ongoing treatment with vitamin K antagonists or oral direct thrombin inhibitors or factor Xa inhibitors (e.g. dabigatran, apixaban or rivaroxaban )
15. Previous arterial bypass surgery (autologous vein or synthetic graft) in the operative leg
16. Stenosis of >50% of the inflow aortoiliac system ipsilateral to the index leg. Any such stenosis must be corrected with angioplasty with or without stenting prior to, or at the time of, HAV implantation
17. Active autoimmune disease - symptomatic or requiring ongoing drug therapy
18. Active local or systemic infection (WBC > 15,000/mm3)
19. Known serious allergy to aspirin
20. Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of the Humacyte Human Acellular Vessel (HAV)
21. Previous exposure to HAV
22. Employees of the sponsor or patients who are employees or relatives of the investigator
23. Pregnant women or women planning to become pregnant (Women of child bearing potential, WOCBP, must use adequate contraception [hormonal or barrier method of birth control; abstinence] for the duration of study participation; WOCBP defined as not sterile or not > 1 year postmenopausal.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shamik Shamik, MD, Study Director — Humacyte, Inc.
Locations (5):
- United States (5):
  - UCSF, San Francisco, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Vascular Center, Flint, Michigan
  - Overlook Medical Center, Summit, New Jersey
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 patients were screened, and 15 patients received the HAV at 6 study centers in the United States of America.
Period: Overall Study
Arm/Group | HAV Treatment
Started | 15
Completed | 0
Not Completed | 15
Not completed — Ongoing | 6
Not completed — Adverse Event | 7
Not completed — Death | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
Age, Customized [Count of Participants; unit: Participants]
  >54 and <75 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (6.00)
Weight [Mean (Standard Deviation); unit: kg] | 81.5 (13.81)
Height [Mean (Standard Deviation); unit: cm] | 168.6 (11.48)
Smoking History [Count of Participants; unit: Participants]
  Former | 11
  Current | 4
  Never | 0
Pack years [Mean (Standard Deviation); unit: Pack years] — One pack-year equals 20 manufactured cigarettes smoked per day for one year
  Pack years | 24.2 (12.46)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Aneurysm Formation, Anastomotic Bleeding or Spontaneous Rupture, HAV Infection, HAV Removal, and Significant Inflammation at the HAV Implantation Site
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
Participants
  Number of Participants with aneurysm formation | 0
  Number of Participants with Anastomotic bleeding or spontaneous rupture | 0
  Number of Participants with HAV infection | 0
  Number of Participants with HAV removal | 0
  Number of Participants with Significant inflammation at the HAV implantation site | 0

2. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
Participants
  Number of Participants with Any AE | 15
  Number of Participants with Mild AEs | 11
  Number of Participants with Moderate AEs | 13
  Number of Participants with Severe AEs | 12
  Number of Participants with Life-threatening AEs | 0
  Number of Participants with Death | 1

3. Primary Outcome: Number of Participants With HAV Patency Rates (Primary, Primary-assisted, Secondary)
Description: Primary patency = patent ("open" to blood flow) without any interventions; Primary-assisted patency = patent without an intervention to clear a thrombus; Secondary patency = patent with or without interventions
Time Frame: 12 months
Population: One patient died prior to the Month 12 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Treatment
Number analyzed (Participants) | 14
Participants
  Number of Participants with Primary Patency at Month 12: Yes | 6
  Number of Participants with Primary Patency at Month 12: No | 8
  Number of Participants with Primary Assisted Patency at Month 12: Yes | 8
  Number of Participants with Primary Assisted Patency at Month 12: No | 6
  Number of Participants with Secondary Patency at Month 12: Yes | 9
  Number of Participants with Secondary Patency at Month 12: No | 5

4. Primary Outcome: Number of Participants With Hemodynamically Significant Stenosis (>70% by Duplex Ultrasound Criteria)
Time Frame: 12 months
Population: One patient did not complete Month 6 visit due to COVID-19-related hospital restrictions; One patient was not assessed at the scheduled Month 9 visit; One patient died prior to the Month 9 visit.
Measure: Number; unit: participants
Arm/Group | HAV Treatment
Number analyzed (Participants) | 14
participants
  Number of Participants with Hemodynamically Significant Stenosis: Month 6 | 2
  Number of Participants with Hemodynamically Significant Stenosis: Month 9: number analyzed (Participants) | 12
  Number of Participants with Hemodynamically Significant Stenosis: Month 9 | 1
  Number of Participants with Hemodynamically Significant Stenosis: Month 12 | 0
  Number of Participants with Hemodynamically Significant Stenosis in Proximal Anastomosis | 2
  Number of Participants with Hemodynamically Significant Stenosis in Distal Anastomosis | 1
  Number of Participants with Hemodynamically Significant Stenosis in Immediate Inflow Artery | 0
  Number of Participants with Hemodynamically Significant Stenosis in HAV Bypass | 0
  Number of Participants with Hemodynamically Significant Stenosis in Immediate Outflow Artery | 0
  Number of Participants with Hemodynamically Significant Stenosis in Presence of Aneurysm | 0

5. Secondary Outcome: Number of Participants With a Change in Panel Reactive Antibodies (PRA) From Baseline
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Treatment
Number analyzed (Participants) | 14
Participants | 0

6. Secondary Outcome: Changes From Baseline in Hematology Parameters - Hemoglobin
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
g/dL
  Hemoglobin (g/dL) | 13.40 (1.69)
  Hemoglobin (g/dL) Change From Baseline | 0.07 (1.24)

7. Secondary Outcome: Changes From Baseline in Coagulation Parameters - International Normalized Ratio (INR)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
ratio
  International Normalized Ratio (INR) | 0.983 (0.067)
  INR Change From Baseline | -0.080 (0.094)

8. Secondary Outcome: Changes From Baseline in Clinical Chemistry Parameters - Sodium, Potassium
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
mmol/L
  Sodium (mmol/L) | 138.3 (3.6)
  Sodium (mmol/L) Change From Baseline | -0.1 (2.0)
  Potassium (mmol/L) | 4.51 (0.34)
  Potassium (mmol/L) Change From Baseline | 0.25 (0.32)

9. Secondary Outcome: Number of Participants With HAV Interventions
Description: e.g., angioplasty, thrombectomy, surgical revision
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
participants
  Number of Participants with HAV intervention due to anastomotic or mid-HAV stenosis | 2
  NUmber of Participant with HAV intervention proximal to the HAV to treat arterial inflow obstruction | 1

10. Secondary Outcome: Mean Vascular Quality of Life Questionnaire (VascuQoL) Score (1-7) for Patients With PAD Symptoms
Description: scoring per Vascular Quality of Life Questionnaire (VascuQoL) Likert scale: 7, there is 1 (the worst) to 7 (the best possible)
Time Frame: 12 months
Population: Mean total VascuQol score at 12 months. One patient died prior to the Month 12 visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HAV Treatment
Number analyzed (Participants) | 14
score on a scale | 5.9 (1.03)

11. Secondary Outcome: Ankle Brachial Index (ABI)
Description: Normal: 1.0 - 1.4 Borderline: 0.9 - 1.0 Mild PAD (peripheral artery disease): 0.8 - 0.9 Moderate PAD: 0.4 - 0.7 Severe PAD: < 0.4
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
units on a scale | 0.902 (0.150)

12. Secondary Outcome: Six Minute Walk Test - Duration
Time Frame: 12 months
Population: One patient did not complete the test. One patient died prior to the Month 12 visit.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
minutes
  Duration (Minutes): number analyzed (Participants) | 13
  Duration (Minutes) | 6.0 (0)
  Change in Duration From Baseline: number analyzed (Participants) | 13
  Change in Duration From Baseline | 0.472 (1.154)

13. Secondary Outcome: Changes From Baseline in Hematology Parameters - Hematocrit
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
percentage
  Hematocrit (%) | 41.69 (4.65)
  Hematocrit (%) Change From Baseline | 1.20 (3.78)

14. Secondary Outcome: Changes From Baseline in Hematology Parameters - Lymphocytes, Monocyte, Eosinophil, Basophil, White Blood Cell, and Neutrophil Counts
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cells x 10^3/uL
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
cells x 10^3/uL
  Absolute Lymphocytes Count (x 10^3/uL) | 2.459 (0.931)
  Absolute Lymphocytes Count (x 10^3/uL) Change From Baseline | -0.186 (0.450)
  Absolute Monocytes Count (x 10^3/uL) | 0.623 (0.133)
  Absolute Monocytes Count (x 10^3/uL) Change From Baseline | 0.004 (0.207)
  Absolute Eosinophils Count (x 10^3/uL) | 0.257 (0.210)
  Absolute Eosinophils Count (x 10^3/uL) Change From Baseline | 0.073 (0.139)
  Absolute Basophils Count (x 10^3/uL) | 0.046 (0.017)
  Absolute Basophils Count (x 10^3/uL) Change From Baseline | 0.009 (0.012)
  White Blood Cells (x 10^3/uL) | 8.399 (2.545)
  White Blood Cells (x 10^3/uL) Change From Baseline | -0.212 (2.103)
  Absolute Neutrophils Count (x 10^3/uL) | 5.079 (1.690)
  Absolute Neutrophils Count (x 10^3/uL) Change From Baseline | 0.046 (1.725)

15. Secondary Outcome: Changes From Baseline in Coagulation Parameters - Activated Partial Thromboplastin Time
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
seconds
  Activated Partial Thromboplastin Time (sec) | 27.26 (3.54)
  Activated Partial Thromboplastin Time (sec) Change From Baseline | 0.18 (2.14)

16. Secondary Outcome: Changes From Baseline in Clinical Chemistry Parameters - Calcium, BUN, Bilirubin, Creatinine, Glucose
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
mg/dL
  Calcium (mg/dL) | 9.38 (0.43)
  Calcium (mg/dL) Change From Baseline | 0.28 (0.51)
  BUN (mg/dL) | 20.9 (17.2)
  BUN (mg/dL) Change From Baseline | 8.7 (16.3)
  Total Bilirubin (mg/dL) | 0.51 (0.21)
  Total Bilirubin (mg/dL) Change From Baseline | -0.02 (0.25)
  Creatinine (mg/dL) | 1.118 (0.471)
  Creatinine (mg/dL) Change From Baseline | 0.188 (0.429)
  Glucose (non-fasting) (mg/dL) | 110.1 (44.2)
  Glucose (non-fasting) (mg/dL) Change From Baseline | 0.9 (29.6)

17. Secondary Outcome: Changes From Baseline in Clinical Chemistry Parameters - Albumin
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
g/dL
  Albumin (g/dL) | 3.93 (0.29)
  Albumin (g/dL) Change From Baseline | 0.39 (0.80)

18. Secondary Outcome: Six Minute Walk Test - Distance
Time Frame: 12 months
Population: One patient did not complete the test. One patient died prior to the Month 12 visit.
Measure: Mean (Standard Deviation); unit: inch
Arm/Group | HAV Treatment
Number analyzed (Participants) | 15
inch
  Distance (in): number analyzed (Participants) | 13
  Distance (in) | 362.514 (143.545)
  Change in Distance From Baseline: number analyzed (Participants) | 13
  Change in Distance From Baseline | 162.049 (164.127)

19. Secondary Outcome: Microscopic Evidence of HAV Remodeling (Host Cells Within HAV)
Time Frame: 12 months
Population: Removal of the HAV would be applicable if there were an indication (e.g., HAV-related complication) for surgical explantation; in this study there were no HAV-related complications warranting the need for surgical excision/removal.
Arm/Group | HAV Treatment
Number analyzed (Participants) | 0

20. Other Pre Specified Outcome: Patient Survival
Time Frame: 60 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Frequency of HAV Remaining as a Functional Conduit in Situ (With or Without Interventions)
Time Frame: 60 months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Evidence of Aneurysmal Dilatation (Conduit Lumen Diameter >9 mm) or Stenosis of the HAV (>70%) on Routine Clinical US
Time Frame: 60 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | HAV Treatment
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 11/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAV Treatment (N=15)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Impaired healing, Oedema peripheral, Pain, Vascular stent restenosis (General disorders) | 4 (5)
Corona virus infection (Infections and infestations) | 1 (1)
Anastomic stenosis, Arterial bypass stenosis, Arterial bypass thrombosis, continued in description (Injury, poisoning and procedural complications) | 9 (15) — Femur fracture, Incision site hematoma
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pleural effusion, Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Arterial insufficiency (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAV Treatment (N=15)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Angina pectoris, Coronary artery disease (Cardiac disorders) | 2 (2)
Implant site extravasation, Peripheral swelling (General disorders) | 4 (5)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Bronchitis, Diverticulitis, Groin infection, Osteomyelitis, Rhinovirus infection (Infections and infestations) | 4 (7)
Post procedural swelling, Seroma, Vascular pseudoaneurysm thrombosis, Wound decomposition (Injury, poisoning and procedural complications) | 2 (2)
Pulse absent, Scan myocardial perfusion abnormal (Investigations) | 2 (2)
Gout, Hyperuricaemia, Vitamin B12 deficiency (Metabolism and nutrition disorders) | 3 (3)
Arthralgia, Back pain, Muscle necrosis, Musculoskeletal pain, Pain in extremity, Tenosynovitis (Musculoskeletal and connective tissue disorders) | 10 (12)
Dizziness, Headache, Neuralgia (Nervous system disorders) | 3 (3)
Anxiety, Insomnia (Psychiatric disorders) | 2 (2)
Renal cyst (Renal and urinary disorders) | 1 (1)
Cough, Pleural effusion, Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dermatitis, Skin hyperpigmentation, Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3)
Arterial stenosis, Haematoma, Intermittent claudication, Continued in description (Vascular disorders) | 9 (13) — Lymphoedema, Peripheral artery dissection, Peripheral artery stenosis, Varicose vein

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and can extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT02887859/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT02887859/SAP_001.pdf